CLINICAL TRIAL: NCT01438372
Title: Intravenous Iron Sucrose Versus Oral Ferrous Sulfate in Treating Iron Deficiency Anemia in Pediatric Inflammatory Bowel Disease
Brief Title: IV Iron Sucrose vs Oral FeSO4 in Treating IDA in Pediatric IBD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated prior to enrolling patients as we were unable to secure enough funding to complete the study.
Sponsor: Wayne State University (Other)
Collaborators: Children's Hospital of Michigan (Other); American Regent, Inc. (Industry)
Responsible Party: Principal Investigator, Mohammad El-Baba, Division Chief, Pediatric Gastroenterology Division, Children's Hospital of Michigan, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1108010039; RR11719 (Other: Detroit Medical Center)
Record Dates: First submitted 2011-09-14; First posted 2011-09-22 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2011-09

CONDITIONS: Iron Deficiency Anemia; Inflammatory Bowel Disease
Keywords: Iron Deficiency Anemia; Inflammatory Bowel Disease; Children
MeSH Terms: conditions — Anemia, Iron-Deficiency; Inflammatory Bowel Diseases | interventions — ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous iron sucrose arm (Experimental)
  Interventions: Drug: Intravenous iron sucrose
- Oral ferrous sulfate (Active Comparator)
  Interventions: Drug: Oral ferrous sulfate

INTERVENTIONS:
Drug: Intravenous iron sucrose — Intravenous iron sucrose will be administered on days 1, 7, 14, and 21 using the formula: Total dose: (normal Hb for age - initial Hb)/100 x blood volume (ml) x 3.4 x 1.5. First dose will be infused over 30 minutes, with subsequent doses administered over 15 minutes if no reactions encountered.
  Other Names: Venofer Luitpold Pharmaceuticals, NDC # 00517-2340-10
  Arms: Intravenous iron sucrose arm
Drug: Oral ferrous sulfate — Oral ferrous sulfate will be administered at 3 mg/kg/day divided into 2 doses for 28 days. A tablet form of ferrous sulfate (325 mg with 65 mg of elemental iron per tablet) will be used.
  Other Names: Upsher-Smith ferrous sulfate 325 mg tablets NDC# 00245-0108-11
  Arms: Oral ferrous sulfate

SUMMARY:
The purpose of this study is to assess the safety and efficacy of intravenous iron sucrose in comparison to oral ferrous sulfate in improving iron deficiency anemia in children with inflammatory bowel disease.

DETAILED DESCRIPTION:
Iron deficiency anemia (IDA) is very common among children with inflammatory bowel disease. Causes in this population are multi-factorial, including decreased absorption due to intestinal disease, increased losses due to bleeding from the gastrointestinal (GI) tract, and poor nutrition. IDA can cause significant impaired physical activity and is associated with developmental and cognitive abnormalities in children and adolescents. Oral ferrous sulfate has been traditionally used to treat iron deficiency anemia, but this is associated with limitations. Studies have shown that only a part of the oral iron is absorbed and the non-absorbed iron salts can be toxic to the intestinal mucosa, and was also theorized to be capable of activating the Inflammatory Bowel Disease (IBD). Use of intravenous iron sucrose has been used in other populations with iron deficiency anemia such as those with chronic kidney disease and children with significant blood loss after spinal surgery. The aim of this study is to determine the safety and efficacy of intravenous iron sucrose in improving iron deficiency anemia in children with inflammatory bowel disease (in comparison to oral ferrous sulfate).

ELIGIBILITY:
Inclusion Criteria:

1. IBD Diagnosis.
2. IDA (defined as a hemoglobin (Hb) concentration of ≤10.5 g/dL females) or Hb ≤11.0 g/dL (males) and Mean Corpuscular volume (MCV) < 77 [22] plus transferrin saturation (TSAT) < 20% and/or serum ferritin concentration less than 25 µg/L)
3. 12- 17 years old males or females.
4. A signed parental permission and assent. Assent is not required in those below 13 years of age.
5. We will be including those who have received iron therapy in the past even if they have developed adverse reactions, as long as they have not been anaphylactic. Participants should have been "iron free" (no iron therapy - oral or IV) for two weeks prior to start of study.

Exclusion Criteria:

1. Anemia other than IDA e.g hemolytic anemia, anemia due to Vitamin B12/Folic acid deficiency.
2. Blood transfusion or iron supplementation 2 two weeks or less before starting the study.
3. Iron overload.
4. Renal disease - on medications such as diuretics or blood pressure lowering medications. On renal replacement therapy.
5. Severe reactive airway disease - classified as severe/high-risk asthma
6. Significant cardiac disease - on cardiac medications, including symptomatic congenital cardiac anomalies or with arrhythmias.
7. Anaphylaxis/hypersensitivity reaction to ferrous sulfate and/or iron sucrose
8. Pregnant and nursing women. A serum pregnancy test will be performed at the start of the study and on days 1, 14, and 28. Patients aged 12 years of age and are found to be pregnant are considered victims of child abuse and will be reported to child protective services and the appropriate authorities.
9. Any other severe concurrent illness.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Safety of IV Iron Sucrose | Up to 56 days
  Safety of IV Iron sucrose is evaluated through timely reporting and thorough description of adverse events. Adverse events related to oral ferrous sulfate will also be reported. Study begins on day of randomization. Iron sucrose is administered on days 1, 7, 14, 21. Follow-up visit is done on day 28 and a follow-up visit or phone call is done on day 49. Oral iron will be taken for 28 days. Patients will be seen in clinic on days 1, 7, 14, 21. With same follow-up as IV iron sucrose.
Efficacy of IV Iron sucrose as measured by change in Hb measurement | baseline and up to 4 weeks.
  Efficacy of IV iron sucrose is evaluated through Hb measurement (gm/dl) at baseline and 4 weeks after treatment with intravenous iron sucrose. (increase of 1 gm/dl in 4 weeks is considered significant). This is compared to Hb increase in participants taking oral ferrous sulfate. Study begins on day of randomization. Iron sucrose is administered on days 1, 7, 14, 21. Follow-up visit is done on day 28 and a follow-up visit or phone call is done on day 49. Oral iron will be taken for 28 days. Patients will be seen in clinic on days 1, 7, 14, 21. With same follow-up as IV iron sucrose.

SECONDARY OUTCOMES:
determine effect on iron parameters: change in transferrin saturation | baseline, and up to 56 days
  would like to determine change in iron parameters: change in transferrin saturation, ferritin levels, serum iron binding capacity. Study begins on day of randomization. Participants have been identified approximately a week before. Iron sucrose is administered on days 1, 7, 14, 21. Follow-up visit is done on day 28 and a follow-up visit or phone call is done on day 49. Oral iron will be taken for 28 days. Patients will be seen in clinic on days 1, 7, 14, 21. With same follow-up as IV iron sucrose.
clinical disease activity | baseline up to 56 days
  to evaluate effects of oral FeSO4 and IV iron sucrose on clinical disease activity. Crohns disease activity will be measured by the Pediatric Crohns Disease Activity Index. Ulcerative colitis disease activity will be measured by Truelove and Witt's classification of severity of ulcerative colitis. Both will be measured at baseline and at 4 weeks. Iron sucrose is administered on days 1, 7, 14, 21. F/u visit is done on day 28 and a f/u visit or phone call is done on day 49. Oral iron will be taken for 28 days. Pts will be seen in clinic on days 1, 7, 14, 21.Same f/u as iron sucrose.
determine effect on iron parameters: change in ferritin levels | baseline up to 56 days
  would like to determine change in iron parameters: change in transferrin saturation, ferritin levels, serum iron binding capacity. Study begins on day of randomization. Participants have been identified approximately a week before. Iron sucrose is administered on days 1, 7, 14, 21. Follow-up visit is done on day 28 and a follow-up visit or phone call is done on day 49. Oral iron will be taken for 28 days. Patients will be seen in clinic on days 1, 7, 14, 21. With same follow-up as IV iron sucrose.
determine effect on iron parameters: change in serum iron binding capacity | baseline up to 56 days
  would like to determine change in iron parameters: change in transferrin saturation, ferritin levels, serum iron binding capacity. Study begins on day of randomization. Participants have been identified approximately a week before. Iron sucrose is administered on days 1, 7, 14, 21. Follow-up visit is done on day 28 and a follow-up visit or phone call is done on day 49. Oral iron will be taken for 28 days. Patients will be seen in clinic on days 1, 7, 14, 21. With same follow-up as IV iron sucrose.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad F El-baba, MD, Principal Investigator — Wayne State University
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States